CLINICAL TRIAL: NCT02783586
Title: Ultrasound Guided Transversus Abdominalis Plane Block ( TAPB) Versus Quadratus Lumborum Type II Block (QLBII) in Perioperative Analgesia for Kidney Transplantation Procedure: Clinical Randomized Multicenter Study
Brief Title: TAPB vs QLBII for Kidney Transplantation Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Kołacz, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAPB/QLB-WAW/OLS
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadratus Lumborum Block type II (Experimental): Unilateral ultrasound guidance QLB on the operated side after induction of general anaesthesia - 20 ml of 0,25%bupivacaine with adrenaline injected with ultraplex needle
  Interventions: Procedure: Quadratus Lumborum Block type II; Drug: Bupivacaine; Device: Ultraplex
- Transversus Abdominalis Plane Block (Active Comparator): Unilateral ultrasound guidance TAPB on the operated side after induction of general anaesthesia - 20 ml of 0,25% bupivacaine with adrenaline injected with ultraplex needle
  Interventions: Procedure: Transversus Abdominalis Plane Block; Drug: Bupivacaine; Device: Ultraplex

INTERVENTIONS:
Procedure: Quadratus Lumborum Block type II — Local anaesthetic injection on the posterior border of the quadratus lumborum muscle
  Arms: Quadratus Lumborum Block type II
Procedure: Transversus Abdominalis Plane Block — Local anaesthetic injection between internal oblique and transversus abdominis muscle
  Arms: Transversus Abdominalis Plane Block
Drug: Bupivacaine — 20 ml of bupivacaine with adrenaline
  Other Names: Marcaine
Device: Ultraplex — A non-stimulating echogenic single-shot needle designed for regional analgesia under ultrasound guidance.

SUMMARY:
The main advantage of Quadratus Lumborum Block (QLB) compared to Transversus Abdominalis Plane Block (TAPB) is the impact on visceral pain due to the spread of the local anaesthetic agent to the paravertebral space. It may produce extensive analgesia and better pain control.

Previews studies shoved the effectiveness of TAPB in kidney transplantation procedure (KTX) by reducing opioids requirements during and after the operation. QLB was not evaluating in KTX procedure yet, but it reduced postoperative morphine requirement after cesarean section under spinal anaesthesia.

The aim of this prospective, randomised controlled, multicenter, clinical study is to compare the perioperative analgesic efficacy of QLB and TAPB in patients who had KTX under balanced (general and regional) anaesthesia.

DETAILED DESCRIPTION:
After Bioethical Committee of Medical University of Warsaw approval, informed written consent will be obtained from all patients.

A sample size of 104 patients was calculated to obtain at list 25% reduction of fentanyl usage in QLBII group with 0,05% significance and power of 0,8. Consenting patients, scheduled to KTX procedure under general anaesthesia will be randomly assigned (1:1) according to the computer -generated randomization list with permuted blocks (block sizes: 20, 20, 24, 40) to receive 20ml of 0,25% Bupivacaine with epinephrine ipsilaterally to the operation side in QLBII or TAPB after the general anaesthesia induction and before the surgery starts. All the blocks will be performed in the supine patients position, under ultrasound guidance for both techniques. The correct spread of injectate will be confirmed with ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplantation procedure with anatomical urinary outlet
2. Written informed consent

Exclusion Criteria:

1. Patients' refusal
2. Known allergies to study medication
3. Inability to comprehend or participate in pain scoring scale
4. Inability to use intravenous patient controlled analgesia system
5. Anatomic, posttraumatic and postoperative deformations could possibly affect the spread of local anesthetic in transversus abdominalis plane or quadratus lumborum muscle plane.
6. Transversus abdominalis plane or quadratus lumborum muscle plane not seen in ultrasound examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Total postoperative fentanyl usage | 24 hours
  Total cumulative fentanyl dose used in the first 24 hours after surgery

SECONDARY OUTCOMES:
Time to first analgesic (TTFA) | 24 hours
  Time from the end of surgery to the first postoperative intravenous fentanyl administered from intravenous patient controlled analgesia ( IVPCA) device.
Postoperative pain severity in Numerical Rating Scale (NRS) in the first 24 hours after surgery | 24 hours
  NRS range from 0 for no pain to 10 for worst pain imaginable.
Nausea or vomiting | 24 hours
  0- no nausea; 1- mild nausea; 2- moderate nausea; 3- severe nausea or vomiting
Sedation Level | 24 hours
  1 - responds to normal verbal communication; 2 - drowsy, but responds to verbal communication; 3- asleep, but awakes with verbal communication; 4- asleep, awakens with mild physical stimulation. 5- asleep, unresponsive to physical stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Kolacz, MD,PhD, Study Director — Medical University of Warsaw; Marcin Mieszkowski, MD, Principal Investigator — Faculty of Medical Sciences, University of Warmia and Mazury in Olsztyn, Poland
Locations (1):
- I Department of Anaesthesiology and Intensive Care, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolacz M, Mieszkowski M, Janiak M, Zagorski K, Byszewska B, Weryk-Dysko M, Onichimowski D, Trzebicki J. Transversus abdominis plane block versus quadratus lumborum block type 2 for analgesia in renal transplantation: A randomised trial. Eur J Anaesthesiol. 2020 Sep;37(9):773-789. doi: 10.1097/EJA.0000000000001193. PMID 32175985